CLINICAL TRIAL: NCT01819948
Title: Pilot Clinical Trial to Assess Changes in Biomarkers of Cancer Related to Inflammation in Women With Stage 0-IIIA Breast Cancer and Without Evidence of Disease Who Were Given the PhytoMed™ Complement.
Brief Title: Changes in Biomarkers of Cancer in Women With Breast Cancer and Without Evidence of Disease Who Were Given PhytoMed™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phytogen Medical Foods S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Phytomed
Record Dates: First submitted 2013-03-13; First posted 2013-03-28 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Stage 0-IIIA; No evidence of disease
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single-arm (Experimental): Two capsules in the morning, one at night, every day for a month, taken with a glass of water.
  Interventions: Dietary Supplement: PhytoMed™

INTERVENTIONS:
Dietary Supplement: PhytoMed™

SUMMARY:
The purpose of this study is to determine whether the administration of the PhytoMed™ complement reduces CRP in women with histologically confirmed AJCC Stage 0-IIIA breast cancer which has been completely surgically resected and without evidence of disease as determined by their physician

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically confirmed AJCC Stage 0-IIIA breast cancer which has been completely surgically resected.
* No evidence of disease as determined by their physician.
* ER+ and/or PR+ tumour.
* Receiving an aromatase inhibitor (letrozole, anastrazole, exemestane) or tamoxifen at a stable dose for at least 3 months at trial entry.
* Post-menopausal women, defined as: (1) above 50 years of age who have not menstruated during the preceding 12 months or who have follicle-stimulating hormone levels (FSH) > 40 IU/L, (2) those under 50 years of age who have FSH hormone levels >40 IU/L, or (3) those who have undergone a bilateral oophorectomy.
* CRP ≥3.9 mg/L measured as the mean of two consecutive weekly tests.
* Aged 18 years or older
* ECOG performance status 0-1
* Between 2 and 5 years from their initial surgery for breast cancer.
* Life expectancy of at least 6 months
* At least 6 months since last chemotherapy
* Laboratory tests performed within 14 days of trial starting:

  1. Granulocytes ≥ 1,500/µL;
  2. Platelets ≥ 100,000/µL;
  3. Haemoglobin ≥ 12.0 g/dL;
  4. Total bilirubin equal to or below upper limit of normal (ULN);
  5. AST and ALT equal to or below ULN;
  6. Alkaline phosphatase equal to or below ULN;
  7. Serum creatinine equal to or below ULN;
* Able to provide informed consent to receive the trial treatment, to provide biological specimens, self-administer oral medica-tion unsupervised for a prolonged period of time, and to complete a medication diary.

Exclusion Criteria:

* Pregnancy or breastfeeding
* Who have had a malignancy (other than breast cancer) which required radiotherapy or systemic treatment within the past 5 years.
* Known cardiac disease (arrhythmias, myocardial infarction, bundle branch block, ischemic heart disease, uncontrolled hypertension)
* Known autoimmune disease or inflammatory disorder
* Any condition requiring the use of systemic corticosteroids or any other immunosuppressive agents (e.g. cyclosporin, tacrolimus, azathioprine).
* Women with known immunodeficiency (such as HIV).
* Patients with infection by septicaemia, infection, acute hepatitis, or other uncontrolled severe medical condition
* Routine use of aspirin >81 mg/d or NSAIDs (> 400 mg po 4 times/day of ibuprofen or naproxen > 500 mg/d) or any use of celecoxib or similar COX-2 inhibitors;
* Subjects are asked not to take dietary supplements, olives or olive oil for 1 month prior to trial enrolment and during the trial.
* Who are taking bisphosphonates

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-06; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Reduction in the levels of CRP | Baseline and 33 +/- 2 days
  Reduction in serum levels of CRP from selection period to end-of-treatment

SECONDARY OUTCOMES:
Reduction in IL-6 | Baseline and 33 +/- 2 days
  Reduction in serum levels of IL-6 from selection period to end-of-treatment
Increase in the levels of IL-10 | Baseline and 33 +/- 2 days
  Increase in serum levels of IL-10 from selection period to end-of-treatment
Safety and tolerability (Gastrointestinal symptoms) | Baseline and 33 +/- 2 days
  Frequency of gastrointestinal adverse events and frequency of patients with gastrointestinal adverse events.
Pain intensity score measured with the BPI scale | Baseline and 33 +/- 2 days
  Pain reduction from selection period to end-of-treatment
Effect on lipid profile | Baseline and 33 +/- 2 days
  Changes in lipid profile from selection period to end-of-treatment
Reduction SAA (serum amyloid A) | Baseline and 33 +/- 2 days
  Reduction in serum levels of SAA from selection period to end-of-treatment
Reduction IFNgamma | Baseline and 33 +/- 2 days
  Reduction in serum levels of IFN gamma from selection period to end-of-treatment
Reduction TNF-alpha | Baseline and 33 +/- 2 days
  Reduction in serum levels of TNF-alpha from selection period to end-of-treatment
Increase in the levels of TGFbeta (transforming growth factor beta) | Baseline and 33 +/- 2 days
  Increase in serum levels of TGF beta from selection period to end-of-treatment
Reduction in IGF (insulin growth factor) | Baseline and 33 +/- 2 days
  Reduction in serum levels of IGF from selection period to end-of-treatment

OTHER OUTCOMES:
Adverse Events | Form start of treatment to day 60
  Frequency and intensity of adverse events and frequency of patients with each adverse event.
Toxicity | Form start of treatment to day 60
  Frequency and intensity of treatment related adverse events and frequency of patients with each treatment related adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Muñoz, Study Chair — Phytogen Medical Foods S.L.
Locations (5):
- Spain (5):
  - Hospital Quirón, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - MD Anderson Cancer Center, Madrid, Madrid